CLINICAL TRIAL: NCT03701308
Title: A Randomized Phase II/III Study of Conventional Chemotherapy +/- Uproleselan (GMI-1271) in Older Adults With Acute Myeloid Leukemia Receiving Intensive Induction Chemotherapy
Brief Title: Daunorubicin and Cytarabine With or Without Uproleselan in Treating Older Adult Patients With Acute Myeloid Leukemia Receiving Intensive Induction Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02130; NCI-2018-02130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A041701 (Other: Alliance for Clinical Trials in Oncology); A041701 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Cytarabine; Daunorubicin; uproleselan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (daunorubicin, cytarabine) (Active Comparator): INDUCTION: Patients receive daunorubicin IV on days 1-3 and cytarabine via CIVI over 168 hours on days 1-7. Patients with residual disease indicated by bone marrow examination receive a second induction including daunorubicin IV on days 1-2 and cytarabine CIVI over 12 hours on days 1-5.
  CONSOLIDATION: Patients receive cytarabine IV over 3 hours on days 1-5. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Additionally, all patients undergo MUGA or ECHO during baseline, and bone marrow aspirate, bone marrow biopsy, and blood collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Arm II (uproleselan, daunorubicin, cytarabine) (Experimental): INDUCTION: Patients receive uproleselan IV QD on day 1 and then every 12 hours on days 2-10. Patients also receive daunorubicin IV on days 2-4 and cytrarabine CIVI over 168 hours on days 2-8 over 168 hours. Patients with residual disease indicated by bone marrow examination receive a second induction including uprleselan IV QD on day 1 and then every 12 hours on days 2-8, daunorubicin IV on days 2-3, and cytarabine CIVI over 120 hours on days 2-6.
  CONSOLIDATION: Patients who achieve a CR or CRi receive uproleselan IV QD on day 1 and every 12 hours on days 2-8 and cytarabine IV over 3 hours on days 2-6. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Additionally, all patients undergo MUGA or ECHO during baseline, and bone marrow aspirate, bone marrow biopsy, and blood collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Uproleselan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Uproleselan — Given IV
  Other Names: GMI-1271
  Arms: Arm II (uproleselan, daunorubicin, cytarabine)

SUMMARY:
This phase II/III trial studies how well daunorubicin and cytarabine with or without uproleselan works in treating older adult patients with acute myeloid leukemia receiving intensive induction chemotherapy. Drugs used in chemotherapy, such as daunorubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Uproleselan may prevent cancer from returning or getting worse. Giving daunorubicin and cytarabine with uproleselan may work better in treating patients with acute myeloid leukemia compared to daunorubicin and cytarabine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the event-free survival (EFS) of daunorubicin, cytarabine plus uproleselan versus daunorubicin and cytarabine in subjects >= age 60 with previously untreated acute myeloid leukemia. (Phase II) II. Compare the overall survival (OS) of the daunorubicin, cytarabine plus uproleselan to daunorubicin and cytarabine in this patient population. (Phase III)

SECONDARY OBJECTIVES:

I. Determine the rates of complete remission (CR), complete remission with incomplete count recovery (CRi), complete remission with incomplete hematopoietic recovery (CRh) and cytogenetic complete remission (CCyR) for each chemotherapy regimen.

II. Determine the overall survival (OS), and remission duration of patients for each chemotherapy regimen.

III. Describe the frequency and severity of adverse events for patients for each chemotherapy regimen.

IV. Describe the interaction of pretreatment disease and patient characteristics including morphology, cytogenetics, molecular genetic features, white blood cell (WBC) count and hemogram, and performance status on clinical outcomes.

CORRELATIVE SCIENCE OBJECTIVES:

I. Correlate specific karyotype groups (normal or various primary and secondary chromosomal abnormalities) with clinical and laboratory parameters and with response rates, response duration, survival and cure in patients treated with various induction and post-induction regimens.

II. Correlate specific karyotype groups with selected molecular abnormalities and with measurable residual disease.

III. To determine karyotype changes at end of consolidation and the influence of the type of change (or no change) in karyotype at the end of consolidation on subsequent clinical course.

IV. To determine karyotype changes at relapse and the influence of the type of change (or no change) in karyotype at relapse on subsequent clinical course.

OUTLINE: Patients are randomized to 1 of 2 arms. (PHASE III CLOSED TO ACCRUAL 08/12/2024)

ARM 1: INDUCTION: Patients receive daunorubicin intravenously (IV) on days 1-3 and cytarabine via continuous intravenous infusion (CIVI) over 168 hours on days 1-7. Patients with residual disease indicated by bone marrow examination receive a second induction including daunorubicin IV on days 1-2 and cytarabine CIVI over 12 hours on days 1-5.

CONSOLIDATION: Patients receive cytarabine IV over 3 hours on days 1-5. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM 2: INDUCTION: Patients receive uproleselan IV QD on day 1 and then every 12 hours on days 2-10. Patients also receive daunorubicin IV on days 2-4 and cytrarabine CIVI over 168 hours on days 2-8 over 168 hours. Patients with residual disease indicated by bone marrow examination receive a second induction including uprleselan IV QD on day 1 and then every 12 hours on days 2-8, daunorubicin IV on days 2-3, and cytarabine CIVI over 120 hours on days 2-6.

CONSOLIDATION: Patients who achieve a CR or CRi receive uproleselan IV QD on day 1 and every 12 hours on days 2-8 and cytarabine IV over 3 hours on days 2-6. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo multigated acquisition scan (MUGA) or echocardiogram (ECHO) during baseline, and bone marrow aspirate, bone marrow biopsy, and blood collection throughout the study.

After completion of study treatment, patients are followed up every 2 months for 1 year, every 3 months in year 2, and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) based on 2017 World Health Organization (WHO) criteria excluding acute promyelocytic leukemia with PML-RARA.

  * Note: Patients with myeloid sarcoma without bone marrow involvement, acute leukemia of ambiguous lineage or blast transformation of chronic myelogenous leukemia (CML) are not eligible.
* No activating mutation in the Fms-like tyrosine kinase-3 (FLT3) defined as a ratio of mutant to wild-type allele >= 0.05 by capillary electrophoresis or a variant allele fraction of >= 5% by next generation sequencing from either bone marrow or peripheral blood.
* No evidence of central nervous system (CNS) involvement of AML.
* No prior chemotherapy for myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN) or AML including hypomethylating agents (e.g. azacitidine and decitabine), ruxolitinib or lenalidomide with the following exceptions:

  * Emergency leukapheresis
  * Hydroxyurea
  * Growth factor/cytokine support
  * All-trans retinoic acid (ATRA)
  * Single dose of intrathecal cytarabine and/or methotrexate for patients undergoing lumbar puncture to evaluate for CNS involvement.
* Age >= 60 years.
* Total bilirubin =< 3 x upper limit of normal (ULN)
* Creatinine < 3 x upper limit of normal (ULN) OR creatinine clearance >= 30 mL/min/1.73m^2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2026-10-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L Uy, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (188):
- United States (188):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Community Cancer Institute, Clovis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Uproleselan, Daunorubicin, Cytarabine): INDUCTION: Patients receive uproleselan IV QD on day 1 and then every 12 hours on days 2-10. Patients also receive daunorubicin IV on days 2-4 and cytrarabine CIVI over 168 hours on days 2-8 over 168 hours. Patients with residual disease indicated by bone marrow examination receive a second induction including uprleselan IV QD on day 1 and then every 12 hours on days 2-8, daunorubicin IV on days 2-3, and cytarabine CIVI over 120 hours on days 2-6.CONSOLIDATION: Patients who achieve a CR or CRi receive uproleselan IV QD on day 1 and every 12 hours on days 2-8 and cytarabine IV over 3 hours on days 2-6. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Additionally, all patients undergo MUGA or ECHO during baseline, and bone marrow aspirate, bone marrow biopsy, and blood collection throughout the study.
Period: Overall Study
Arm/Group | Arm I (Daunorubicin, Cytarabine) | Arm II (Uproleselan, Daunorubicin, Cytarabine)
Started | 136 | 131
Completed | 134 | 129
Not Completed | 2 | 2
Not completed — Ineligible | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Daunorubicin, Cytarabine) | Arm II (Uproleselan, Daunorubicin, Cytarabine) | Total
Number analyzed (Participants) | 136 | 131 | 267
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.1 [63.8 to 69.9] | 66.8 [63.6 to 69.9] | 66.9 [63.8 to 69.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 60 | 110
  Male | 86 | 71 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 121 | 109 | 230
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 12 | 22
  White | 119 | 99 | 218
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 5 | 17 | 22

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the time from the date of randomization to the first of failure to achieve a complete remission (CR)/ CR with incomplete blood count recovery (CRi) during induction, relapse, or death due to any cause, with patients last known to be alive and event-free censored at the date of last contact.
Time Frame: 67 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Daunorubicin, Cytarabine) | Arm II (Uproleselan, Daunorubicin, Cytarabine)
Number analyzed (Participants) | 134 | 129
months | 5.4 [3.3 to 8.3] | 9.4 [5.2 to 13.8]

2. Primary Outcome: Overall Survival (OS)
Description: Will be measured from the date of randomization to death from any cause, with patients last known to be alive censored at the date of last contact.
Time Frame: 67 months
Population: All registered patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Daunorubicin, Cytarabine) | Arm II (Uproleselan, Daunorubicin, Cytarabine)
Number analyzed (Participants) | 136 | 131
Months | 19.8 [14.6 to 43.3] | 23.6 [15.1 to 35.3]

3. Secondary Outcome: EFS Rate at 24 Months
Description: Event Free Survival will be defined as the time from patient registration to treatment failure, progression, or death. The proportion of patients alive and event free at 24 months will be reported.
Time Frame: 24 months
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Arm I (Daunorubicin, Cytarabine) | Arm II (Uproleselan, Daunorubicin, Cytarabine)
Number analyzed (Participants) | 134 | 129
proportion of patients | 0.290 [0.215 to 0.390] | 0.326 [0.249 to 0.426]

4. Secondary Outcome: Impact of Off-protocol Transplantation
Description: Sensitivity analyses will be conducted. In addition, the proportion of patients who received transplantation in the two arms will be summarized and compared using a chi-square test.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Consistency of the Treatment Effect Among Each Subgroup
Description: Non-parametric methods such as Kaplan-Meier and log-rank tests will be used within each subgroup. Univariate/multivariate Cox models will be fit within each subgroups; hazard ratios will be used to quantify the treatment effect within each subgroup, along with the 95% confidence intervals.
Time Frame: From baseline up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Disease-free Survival (DFS)
Time Frame: Time from achieving a complete response to time of relapse or death, assessed up to 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Complete Remission (CR) and Overall Response Rate
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 5.0. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Prediction of CR, EFS, DFS, and OS by Pretreatment Characteristics Such as Age, Morphology, Cytogenetics, Immunophenotype, Molecular Genetic Features, WBC Count and Hemogram, and Performance Status With Clinical Outcomes
Description: The associations between these baseline factors and CR, EFS, DFS, and OS will be analyzed using Kaplan-Meier curves, log-rank test, contingency table and chi-square test whenever appropriate. Multivariable analysis including Cox proportional hazards models and logistic regression models will be used as well to evaluate the associations.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 25 months and mortality was followed for 67 months.
Arm/Group | Arm I (Daunorubicin, Cytarabine) | Arm II (Uproleselan, Daunorubicin, Cytarabine)
All-Cause Mortality (participants affected / at risk) | 47/136 | 84/131
Serious Adverse Events (participants affected / at risk) | 12/136 | 12/131
Other Adverse Events (participants affected / at risk) | 130/136 | 126/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Daunorubicin, Cytarabine) (N=136) | Arm II (Uproleselan, Daunorubicin, Cytarabine) (N=131)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 4 (4)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Daunorubicin, Cytarabine) (N=136) | Arm II (Uproleselan, Daunorubicin, Cytarabine) (N=131)
Anemia (Blood and lymphatic system disorders) | 99 (359) | 103 (405)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 3 (4) | 2 (9)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 107 (137) | 95 (149)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (8) | 11 (14)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (2) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 2 (2)
Heart failure (Cardiac disorders) | 4 (6) | 1 (3)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 8 (9)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 4 (5) | 3 (3)
Eye pain (Eye disorders) | 1 (1) | 2 (2)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (2) | 0 (0)
Periorbital edema (Eye disorders) | 2 (2) | 1 (1)
Vision decreased (Eye disorders) | 2 (2) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 20 (21) | 11 (13)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (3)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 28 (36) | 22 (32)
Dental caries (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 83 (117) | 79 (119)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 9 (12)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (8) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 4 (4) | 4 (8)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (3) | 4 (5)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 47 (78) | 50 (72)
Nausea (Gastrointestinal disorders) | 81 (128) | 81 (154)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4)
Oral pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Proctitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 4 (6) | 3 (4)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 4 (5)
Typhlitis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (15) | 14 (21)
Chills (General disorders) | 9 (13) | 9 (10)
Edema face (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 12 (17) | 23 (27)
Fatigue (General disorders) | 46 (73) | 48 (85)
Fever (General disorders) | 20 (25) | 24 (35)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 7 (30) | 8 (21)
Generalized edema (General disorders) | 3 (3) | 4 (8)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 2 (4) | 5 (7)
Malaise (General disorders) | 3 (4) | 7 (8)
Non-cardiac chest pain (General disorders) | 3 (3) | 6 (6)
Pain (General disorders) | 3 (3) | 8 (12)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2) | 3 (3)
Abdominal infection (Infections and infestations) | 3 (3) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 9 (10) | 6 (6)
Bone infection (Infections and infestations) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 6 (7) | 7 (9)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 15 (19) | 20 (32)
Lung infection (Infections and infestations) | 14 (14) | 16 (21)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (2) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 4 (5)
Sepsis (Infections and infestations) | 24 (27) | 19 (24)
Sinusitis (Infections and infestations) | 3 (3) | 4 (5)
Skin infection (Infections and infestations) | 6 (8) | 6 (9)
Thrush (Infections and infestations) | 9 (10) | 4 (5)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 4 (5) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 4 (5)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Activated partial throm time prolonged (Investigations) | 3 (3) | 1 (4)
Alanine aminotransferase increased (Investigations) | 66 (130) | 72 (164)
Alkaline phosphatase increased (Investigations) | 6 (9) | 11 (21)
Aspartate aminotransferase increased (Investigations) | 58 (101) | 67 (126)
Blood bilirubin increased (Investigations) | 53 (95) | 58 (85)
Blood lactate dehydrogenase increased (Investigations) | 3 (5) | 4 (10)
Cardiac troponin I increased (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 12 (18) | 10 (14)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 6 (8) | 3 (6)
Fibrinogen decreased (Investigations) | 0 (0) | 2 (2)
GGT increased (Investigations) | 0 (0) | 2 (4)
INR increased (Investigations) | 6 (7) | 4 (6)
Investigations - Other, specify (Investigations) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 63 (275) | 67 (316)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 84 (332) | 88 (354)
Platelet count decreased (Investigations) | 103 (472) | 110 (508)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 6 (7)
Weight loss (Investigations) | 6 (8) | 11 (19)
White blood cell decreased (Investigations) | 102 (419) | 103 (478)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 26 (34) | 39 (54)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (26) | 19 (31)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 8 (8)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 6 (9) | 11 (12)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 35 (53) | 31 (57)
Hypocalcemia (Metabolism and nutrition disorders) | 29 (44) | 22 (48)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 35 (50) | 34 (65)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (12) | 6 (8)
Hyponatremia (Metabolism and nutrition disorders) | 11 (14) | 10 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (15) | 15 (23)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (4)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 10 (10) | 14 (15)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (5) | 6 (7)
Encephalopathy (Nervous system disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 12 (18) | 25 (35)
Intracranial hemorrhage (Nervous system disorders) | 3 (3) | 4 (4)
Lethargy (Nervous system disorders) | 2 (2) | 3 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Reversbl posterior leukoenceph syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (2) | 2 (2)
Syncope (Nervous system disorders) | 3 (3) | 7 (7)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 7 (9) | 8 (9)
Confusion (Psychiatric disorders) | 4 (4) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 3 (7)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (7) | 11 (13)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (7) | 5 (5)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 1 (1)
Glucosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (4) | 4 (5)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (3)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (4) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 11 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (27) | 22 (24)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 14 (16)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 12 (14)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 10 (12)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (5) | 11 (25)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (26) | 18 (27)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 5 (7) | 9 (21)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 1 (2)
Hematoma (Vascular disorders) | 1 (1) | 3 (4)
Hypertension (Vascular disorders) | 17 (26) | 17 (31)
Hypotension (Vascular disorders) | 20 (25) | 17 (22)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (2)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (10)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 2 (2)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03701308/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03701308/ICF_001.pdf